CLINICAL TRIAL: NCT04628442
Title: Tissue Immune Interaction in Nasal Polyposis
Acronym: TIP
Status: Completed | Type: Observational
Sponsor: University of California, San Francisco (Other)
Collaborators: National Institutes of Health (NIH) (NIH); National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Sponsor
Other Study IDs: 19-28725; 2P01HL107202-06A1 (NIH)
Record Dates: First submitted 2020-02-27; First posted 2020-11-13 (Actual); Last update posted 2025-07-30 (Actual); Status verified 2025-07

CONDITIONS: Chronic Rhinosinusitis (Diagnosis); Chronic Rhinosinusitis With Nasal Polyps; Asthma
Keywords: Asthma; Chronic Rhinosinusitis; Surgery
MeSH Terms: conditions — Disease; Asthma | interventions — Biopsy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — Nasal polyp tissue collected from the nasal passages, inferior turbinate tissue collected form the nasal passages, mucus collected from the nasal passages, induced sputum, and blood.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- TIP-OB (Office-Based): Those in TIP-OB will be undergoing regularly scheduled office-based procedures at the otolaryngology clinic at UCSF Mount Zion campus. The investigators will be collecting nasal mucus and blood samples during each of their visits to the clinic, up to 9 times.
  Interventions: Procedure: Sinonasal Debridement Procedure
- TIP-OR (Operating Room): Those in TIP-OR will be undergoing regularly scheduled surgeries in the operating room at UCSF Parnassus or Mount Zion campus. The investigators will be collected nasal polyp tissue, nasal mucus if possible, and blood samples during each of their surgeries, up to 9 times. The investigators will also collect inferior turbinate tissue if consented to.
  Interventions: Procedure: Nasal Polyp Removal; Procedure: Biopsy

INTERVENTIONS:
Procedure: Sinonasal Debridement Procedure — This is a medical procedure prescribed by the participant's physician that has been deemed necessary for patient care in order to address their chronic rhinosinusitis.
  Groups: TIP-OB (Office-Based)
Procedure: Nasal Polyp Removal — This is a surgical procedure prescribed by the participant's physician that has been deemed necessary for patient care in order to address their chronic rhinosinusitis.
  Groups: TIP-OR (Operating Room)
Procedure: Biopsy — A biopsy is optional and will remove a sample of inferior turbinate tissue from the nasal passage. It will be performed during a nasal polyp removal surgery already scheduled for patient care.
  Groups: TIP-OR (Operating Room)

SUMMARY:
This is a cross-sectional study of up to 100 subjects who are undergoing clinically indicated sinus procedures to treat chronic rhinosinusitis. Participants will be asked to donate leftover sino-nasal secretions, sino-nasal tissue and blood as well as undergo partial characterization. As optional extensions of the main study, participants may also undergo a biopsy of extra sino-nasal tissue for additional tissue analysis and/or a more detailed characterization visit performed in the UCSF Airway Center Research Center (ACRC).

DETAILED DESCRIPTION:
This is a cross-sectional study of up to 100 participants who are undergoing clinically indicated sinus procedures to treat chronic rhinosinusitis. 50 participants with CRSwNP and 50 participants with CRS without polyps and no features of atopy will be enrolled in the study. Participants will donate leftover sino-nasal secretions and tissue from their procedures. In addition, participants will be subject to medical record review and research questionnaires.

In many instances, these participants will have multiple procedures over time to treat recurrent disease and this study will allow for them to donate leftover biospecimens as many as 9 times.

Participants may also opt to undergo a turbinate mucosal tissue biopsy during regularly scheduled sinus surgery for additional tissue analysis and/or undergo a more detailed, complete characterization visit performed in the UCSF Airway Center Research Center (ACRC). During the complete characterization, participants will undergo lung function tests, sputum induction and blood collection, in addition to the procedures mentioned above.

ELIGIBILITY:
Participants with Chronic Rhinosinusitus with Nasal Polyps

Inclusion Criteria:

* Males or females between the ages 18 to 80 (inclusive).
* History of blood eosinophils > 200 cells/dL (or tissue eosinophilia evident on histopathologic review of sino-nasal tissues).
* Physician diagnosis of chronic rhinosinusitis (CRS).
* Undergoing office-based or operating room-based sinus procedures for a clinical indication.
* Written informed consent obtained from subject and ability for subject to comply with the requirements of the study.

Exclusion Criteria:

* Smoking of tobacco or other recreational inhalants more than twice in the last month and/or >10 pack-year smoking history.
* History of cystic fibrosis or ciliary dyskinesia.
* Currently taking immunosuppressant drugs including Mycophenolate mofetil (Cellcept), Cyclophosphamide (Cytoxan), Azathioprine (Imuran).

Participants with Chronic Rhinosinusitus without Nasal Polyps

Inclusion Criteria:

* Males or females between the ages 18 to 80 (inclusive)
* Physician diagnosis of CRS.
* Undergoing office-based or operating room-based sinus procedures for a clinical indication.
* Written informed consent obtained from subject and ability for subject to comply with the requirements of the study.

Exclusion Criteria:

* Smoking of tobacco or other recreational inhalants more than twice in the last month and/or >10 pack-year smoking history.
* Presence of nasal polyps.
* History of allergic rhinitis.
* History of blood eosinophilia > 200 (or tissue eosinophilia evident on histopathologic review of sino-nasal tissues).
* Currently taking immunosuppressant drugs including Mycophenolate mofetil (Cellcept), Cyclophosphamide (Cytoxan), Azathioprine (Imuran).

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Participants with chronic rhinosinusitis who present with or without nasal polyps between the ages of 18 and 80 years.
Sampling Method: Non-Probability Sample
Enrollment: 38 (Actual)
Dates: Start 2020-11-10 (Actual); Primary Completion 2023-03-24 (Actual); Study Completion 2023-03-24 (Actual)

PRIMARY OUTCOMES:
Percentage of ILC2 and tuft cells | Up to 8 hours
  This study enrolls chronic rhinosinusitis patients with and without nasal polyps. Investigators aim to compare the percentage of ILC2 and tuft cells present in nasal tissue and secretions between those who present with nasal polyps and without nasal polyps.

CONTACTS AND LOCATIONS:
Overall Officials: John Fahy, MD, MSc, Principal Investigator — University of California, San Francisco
Locations (1):
- UCSF Airway Clinical Research Center, San Francisco, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Airway Clinical Research Center website — http://acrc.ucsf.edu